CLINICAL TRIAL: NCT03286374
Title: Do Change in Life Style Improve Work Ability? A Controlled Study of the Effect of Changes in Lifestyle on Work Participation.
Brief Title: Do Change in Life Style Improve Work Ability?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Collaborators: Volda University College (Other)
Responsible Party: Principal Investigator, Anita Dyb Linge, Ph.D Student, Molde University College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017/573
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Obesity, Morbid; Sick-leave; Work Related Illnesses; Life Style
Keywords: Obesity; Occupational rehabilitation; Sick leave; Life style treatment
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Intervention Model Description: The study is a Clinical cohort trial with a pseudo prospective, parallel mixed methods design. Questionnaires and register data at baseline, T1, and T2. Focus group interviews at T3, and register data at T4.
Masking Description: Due to the nature of the study intervention, it is not possible to blind the participants. Some of the participants will give a focus group interview and their identity will be known for the other participants in the group. The health care providers will not get information about who will participate or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupational rehabilitation (Other): The participants will receive the current occupational rehabilitation program at Muritunet.
  Interventions: Behavioral: Occupational rehabilitation

INTERVENTIONS:
Behavioral: Occupational rehabilitation — The participants in the occupational rehabilitation program get both practical and theoretical intervention in groups. Four main interventions; cognitive therapy, physical activity, diets and training in work-oriented approach. The rehabilitation stay is as followed:
  1. Four weeks with an institutional stay at Muritunet (BL)
  2. Follow-up;
     1. Eight weeks, telephone contact between therapist at Muritunet and the participant.
     2. 16 weeks, video conference on SKYPE between all the participants and a therapist. Lecture on diets.
     3. 28 weeks, Follow-up at Muritunet. Central themes that day is education, conversation, physical test, and forms. (T1)
     4. 40 weeks, telephone contact between therapist at Muritunet and the participant.
     5. 52 weeks, Follow-up at Muritunet. Central themes that day is education, conversation, physical test, and forms. (T2)
  Other Names: Life style treatment

SUMMARY:
The main aim of this Cohort trial is to get more information about how life style changes affect work participation for people with BMI above 30. The information can contribute to improving the quality of occupational rehabilitation programs in the specialized health care services and for others who work with weight loss programs and work related rehabilitation programs.

DETAILED DESCRIPTION:
The goal of rehabilitation, in general, is to help people to reach and maintain their optimal function and copying capabilities and to promote independence and participation in society. For occupational rehabilitation is the goal also to increase function and work ability to prevent the individuals permanent to fall out of working life. People with high BMI needs beside work rehabilitation also focus on life style changes to reduce consequences of obesity. The Central Norway Regional Health Authority (HMN RHF) has initiated action to reduce work absence and consequence of obesity by introducing a work related rehabilitation program for people with BMI above 30. This program combines work participation and life style changes and exists only in two institutions in Norway. The goal of the program is to increase function and work ability and weight loss. The program is new, and few documents exist on the effect and the correlation between life style changes and work ability. There is also need to question whether obesity is the reason for work absence or is there other factors that affect work ability. This trial wants to follow-up a group of people who have been participating occupational rehabilitation at Muritunet.

ELIGIBILITY:
Inclusion Criteria:

1. People who are on sick leave or stands in danger of being sick because of problems related to obesity.
2. The participants must have a realistic opportunity to return to work.
3. Body mass index above 30
4. Age 18-67 years.

Exclusion criteria;

1. People with a severe eating disorder.
2. People without a capacity to consent.
3. People with severe alcohol and/or drug abuse.
4. People with a major mental illness.
5. Being pregnant.
6. People with a health condition that contraindicates physical activity.
7. People who receive work assessment allowance.
8. People with or plan to apply for disability benefits.
9. People with permanently adapted work.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Work participation | 1-4 years
  Work participation after a work related rehabilitation program at Muritunet.

SECONDARY OUTCOMES:
Life quality | Survey data collected at baseline, six and twelve months after participation in the trial.
  Quality of life; health - 15D ( Harri Sintonen, http://www.15d-instrument.net)
Work motivation | Survey data collected at baseline, six and twelve months after participation in the trial.
  Return to work self-efficacy, Return-to-work self-efficacy scale (RTWSE-19) (Shaw et al. 2011)
Weight loss | Weight collected at baseline, six and twelve months after participation in the trial.
  Weight changing

CONTACTS AND LOCATIONS:
Overall Officials: Odd Ragnar Hunnes, Dean, Study Director — Volda University Collage
Locations (1):
- Anita Dyb Linge, Valldal, Møre og Romsdal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Linge AD, Bjorkly SK, Jensen C, Hasle B. Bandura's Self-Efficacy Model Used to Explore Participants' Experiences of Health, Lifestyle, and Work After Attending a Vocational Rehabilitation Program with Lifestyle Intervention - A Focus Group Study. J Multidiscip Healthc. 2021 Dec 24;14:3533-3548. doi: 10.2147/JMDH.S334620. eCollection 2021. PMID 34992380
- [Derived] Linge AD, Jensen C, Laake P, Bjorkly SK. Changes to body mass index, work self-efficacy, health-related quality of life, and work participation in people with obesity after vocational rehabilitation: a prospective observational study. BMC Public Health. 2021 May 17;21(1):936. doi: 10.1186/s12889-021-10954-y. PMID 34001067

DOCUMENTS (1):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03286374/Prot_000.pdf